CLINICAL TRIAL: NCT03178123
Title: A Phase II Randomized, Control, Multi-center Study of Recombinant Humanized Anti-PD-1 mAb for Injection Compared to High-Dose Interferon In Patients With Mucosal Melanoma That Has Been Removed by Surgery
Brief Title: The Study of JS001 Compared to High-Dose Interferon In Patients With Mucosal Melanoma That Has Been Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Junshi-JS001-010
Record Dates: First submitted 2017-05-27; First posted 2017-06-06 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Mucosal Melanoma
Keywords: anti-PD-1 monoclonal antibody; Mucosal Melanoma; Interferons
MeSH Terms: interventions — Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- humanized anti-PD-1monoclonal antibody (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 3mg/kg Q2w until disease progresses or unacceptable tolerability occurs for 1 year (27 treatments)
  Interventions: Biological: humanized anti-PD-1 monoclonal antibody Toripalimab
- high-dose recombinant interferon a-2B (Active Comparator): Patients receive 15*10^9 U/m2/d recombinant interferon a-2B intravenously on days 1-5. Treatment repeats weekly for 4 weeks in the absence of disease progression or unacceptable toxicity.Then patients receive 15*10^9 U/m2/d recombinant interferon a-2B intravenously three times weekly for 48 weeks.
  Interventions: Biological: high-dose recombinant interferon a-2B

INTERVENTIONS:
Biological: humanized anti-PD-1 monoclonal antibody Toripalimab — humanized anti-PD-1 monoclonal antibody (JS001) is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with the combination of PD-1 with its ligands, PD-L1 and PD-L2, resulting in the activation of lymphocytes and elimination of malignancy theoretically.
  Other Names: JS001, TAB001
  Arms: humanized anti-PD-1monoclonal antibody
Biological: high-dose recombinant interferon a-2B — 15*10^9 U/m2/d recombinant interferon a-2B intravenously on days 1-5 weekly for 4 weeks.Then 15*10^9 U/m2/d recombinant interferon a-2B intravenously three times weekly for 48 weeks.
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Intron A
  Arms: high-dose recombinant interferon a-2B

SUMMARY:
This is a phase II randomized, control, multi-center study of recombinant humanized anti-PD-1 mAb for injection compared to high-Dose interferon in patients with mucosal melanoma that has been removed by surgery.

DETAILED DESCRIPTION:
This is a multi-centre，open, randomized, parallel-group study of mucosal melanoma adjuvant therapy to evaluate the efficacy of recombinant humanized anti-PD-1 mAb for injection compared to high-Dose interferon in patients with mucosal melanoma that has been removed by surgery.There will be 220 subjects enrolling the study, and randomized 1:1 grouped into recombinant humanized anti-PD-1 mAb for injection group (experimental group) or interferon group (control group).Each group will have 110 subjects.Random stratification factor is the disease stage (I vs II vs III).The whole research lasts about 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged between 18 and 75 years are eligible;
* It was confirmed by histopathology that it was a mucosal melanoma;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* Complete excision of primary focal area, surgical incision; All patients must have disease-free status documented by a complete physical examination and imaging studies prior to registration;
* No adjuvant therapy was received;
* No treatment contraindication, peripheral blood, normal liver, kidney function and electrocardiogram are normal; WBC≥4.0×10^9/L,PLT≥100×10^9/L,Hgb≥90g/L; serum urea nitrogen, cr≤ULN; ALT,AST,TBI≤1.5*ULN,
* Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 12 months after the last dose of study drug;
* FT3,FT4 and TSH is normal;
* Must have read, understood, and provided written informed consent voluntarily. Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Prior treatment with anti-PD-1/PD-L1/PD-L2 antibody;
* Hypersensitivity to recombinant humanized anti-PD-1 monoclonal mAb or its components;
* Skin melanoma, ocular melanoma, original unknown melanoma;
* The primary lesion was incomplete;
* The examination suggests that the tumor remains or metastases;
* Pregnant or nursing;Women with fertility but not contraception;
* There are severe acute infections that are not controlled;There is a suppurative and chronic infection, and the wound is deferrable;
* Those who had serious heart disease;
* Psychiatric medicines abuse without withdrawal, or history of psychiatric illness.
* Patients with other tumor;
* Participate in other clinical studies at the same time;
* Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml);
* Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism;
* Prior live vaccine therapy within past 4 weeks;
* Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival rate | 5 years
  to evaluate the Recurrence free survival (RFS) of the patients with mucosal melanoma treated by JS001 and high-Dose interferon

SECONDARY OUTCOMES:
Distant metastases-free survival | 5 years
  to evaluate the distant metastases-free survival of the patients with mucosal melanoma treated by JS001 and high-Dose interferon
recurrence - free survival rate at 3 years | 3 years
  to evaluate the recurrence - free survival rate at 3 years of the patients with mucosal melanoma treated by JS001 and high-Dose interferon
Overall survival (OS) | 5 years
  to evaluate the Overall survival (OS) of the patients with mucosal melanoma treated by JS001 and high-Dose interferon
Number of participants with treatment-related adverse events | 5 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes